CLINICAL TRIAL: NCT03898635
Title: Retrospective Real-word Study of Linezolid for the Treatment of Tuberculous Meningitis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Wen-hong Zhang, Director of Division of Infectious Diseases, Huashan Hospital
Other Study IDs: 2017-44
Record Dates: First submitted 2019-03-28; First posted 2019-04-02 (Actual); Last update posted 2019-04-02 (Actual); Status verified 2019-03

CONDITIONS: Tuberculous Meningitis
Keywords: linezolid
MeSH Terms: conditions — Tuberculosis, Meningeal | interventions — Linezolid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Background group: The treatment regimen does not include linezolid throughout the treatment course.
- Background-linezolid group: Linezolid was added in the middle of the treatment course but not in the initial treatment regimen.
  Interventions: Drug: Linezolid
- Linezolid initial group: Linezolid was in initial treatment regimen.
  Interventions: Drug: Linezolid

INTERVENTIONS:
Drug: Linezolid — To add linezolid 600mg or 1200mg daily in the initial or subsequent treatment regimen of TBM.
  Groups: Background-linezolid group; Linezolid initial group

SUMMARY:
Tuberculous meningitis (TBM) is the most serious form of Mycobacterium tuberculosis infection, causing mortality and disability in more than half of the patients. Current standard treatment for TBM is based on those developed to treat pulmonary tuberculosis, which does not take into account the differential ability of anti-tuberculosis drugs to penetrate the brain. With both good central nervous system penetrance and anti-tuberculosis efficacy that have been demonstrated in drug-resistant tuberculosis, linezolid may be a promising antimicrobial in TBM treatment. The purpose of this study is to evaluate the effectiveness of linezolid in the treatment of TBM.

ELIGIBILITY:
Inclusion Criteria:

* all patients diagnosed as TBM from the electronic medical record system.

Exclusion Criteria:

* Does not meet the established diagnostic criteria;
* Combine other pathogen central infections;
* Follow-up confirmed that the final diagnosis considers other diseases (such as tumors, autoimmune encephalitis, etc.);
* Our hospital has less than one week of anti-tuberculosis treatment;
* Lack of information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with central nervous system tuberculosis diagnosed and treated at Huashan Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-05-01 (Estimated); Study Completion 2019-06-01 (Estimated)

PRIMARY OUTCOMES:
Survival | 5 years

SECONDARY OUTCOMES:
Number of participants with Medical Research Council grade deterioration | From the beginning of anti-tuberculosis treatment to the first documented progression, assessed up to 5 years.

OTHER OUTCOMES:
Time of Glasgow Coma Scale recovered to 15 | From the beginning of anti-tuberculosis treatment to the first documented recovery, assessed up to 5 years.
Time of body temperature returns to normal | From the beginning of anti-tuberculosis treatment to the first documented recovery, assessed up to 5 years.
Number of participants with new omplications | From the beginning of anti-tuberculosis treatment to the first documented progression, assessed up to 5 years.
  Hydrocephalus, cerebral infarction, epilepsy, brain abscess, tuberculoma

CONTACTS AND LOCATIONS:
Locations (1):
- Infectious department of Huashan Hospital, Fudan University, Shanghai, China